CLINICAL TRIAL: NCT00428233
Title: Banking of Chronic Lymphocytic Leukemia Tumor Cells for Vaccine Generation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Catherine Wu, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-200
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; vaccine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Leukemia Cell Harvest (No Intervention): Procedure/Surgery: Leukemia cell harvest Leukemia cells will be harvested either by: Blood draw, leukapheresis, bone marrow aspiration or surgery to remove the lymph node
  Interventions: Procedure: Leukemia cell harvest

INTERVENTIONS:
Procedure: Leukemia cell harvest — Leukemia cells will be harvested either by: Blood draw, leukapheresis, bone marrow aspiration or surgery to remove the lymph node

SUMMARY:
The purpose of this research study is to collect, freeze and store leukemia cells from the blood or bone marrow of patients that have advanced chronic lymphocytic leukemia (CLL) that is not in clinical remission. This study is a companion study to DF/HCC clinical trial 06-196 in which the participants' own CLL cells may form part of a vaccine treatment for their leukemia.

DETAILED DESCRIPTION:
* It is important to understand that even if the participant consents to allow us to save their leukemia cells, we cannot guarantee that they will be able to receive a vaccine. First, we may not be able to make enough vaccine from the collected cells. Second, they may not be able to participate in a vaccine study in the future for reasons related to the status of your overall health. Third, an appropriate vaccine trial may not be available in the future.
* In order to make the vaccine, leukemia cells will be collected by one or more of the following methods: drawing blood during one of two visits to the clinic; leukapheresis; bone marrow aspiration; or, surgery to remove a lymph node.
* The physician will discuss with the participant which approach is best in their case to ensure the highest number of tumor cells collected.

ELIGIBILITY:
Inclusion Criteria:

* Ability to harvest CLL cells from peripheral blood, lymph nodes or bone marrow, defined as > 30% involvement of bone marrow intratrabecular space, or peripheral blood lymphocytosis > 5000/microliter, or surgically accessible lymph nodes of greater than or equal to 2cm.
* ECOG performance status 0-2
* 18 years of age or older

Exclusion Criteria:

* Uncontrolled infection
* Leukemia with active CNS involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To collect up to 20 patient samples per year that could potentially be used to prepare autologous tumor cell vaccines. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J. Wu, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States